CLINICAL TRIAL: NCT06206265
Title: A Phase 2a, Open-label, Pilot Study to Assess the Safety and Efficacy of Oral Psilocybin (TRP-8802) Administration in Concert With Psychotherapy Among Adult Patients With Irritable Bowel Syndrome: A Randomized Delayed Treatment Control Design
Brief Title: Assessment of Psilocybin (TRP-8802) in Concert With Psychotherapy in Patients With Irritable Bowel Syndrome (IBS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TRYP Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRYP-003
Record Dates: First submitted 2023-09-12; First posted 2024-01-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized either into the immediate therapy vs. waitlist control. Patients in the waitlist control will eventually be offered the same therapy at 8 weeks post enrollment. The delayed treatment arm will initiate therapy on the same schedule as the immediate treatment arm.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open Label Oral Psilocybin (Experimental)
  Interventions: Drug: TRYP-0082; Behavioral: Psychotherapy
- Waitlist Control (Other)
  Interventions: Drug: TRYP-0082; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: TRYP-0082 — Participants will receive one dose of 25 mg of oral psilocybin on the first dosing day and a second dose of 25mg oral psilocybin on the second dosing day. TRP 8802 will be administered in a comfortable setting under the guidance of the same two therapists from the preparation period. Participants will have an in-person study visit following the resolution of the psychoactive effects of the psilocybin (as determined by the therapists in discussion with the participant) to ensure participant's safety and comfort.
Behavioral: Psychotherapy — Participants will receive one dose of 25 mg of oral psilocybin on the first dosing day and a second dose of 25mg oral psilocybin on the second dosing day. TRP 8802 will be administered in a comfortable setting under the guidance of the same two therapists from the preparation period. Participants will have an in-person study visit following the resolution of the psychoactive effects of the psilocybin (as determined by the therapists in discussion with the participant) to ensure participant's safety and comfort.

SUMMARY:
Participants with IBS (all subtypes) and with no exclusionary comorbid psychiatric or medical disorders will be enrolled in the study.

This study will involve a randomized waitlist control design to investigate the rapid and sustained effects of TRP-8802 following two experimental sessions in which an oral dose of TRP-8802 is administered to participants with IBS. The study will include clinician and participant ratings of depression and anxiety pre- and post-drug-session, monitor and participant ratings of subjective drug effects during and after each drug session.

This study comprises approximately a 28-day screening period (Days 28 to 1). After screening and enrollment, participants will be randomized to an immediate treatment group or a delayed treatment group ("waitlist control" condition).

Participants in the immediate treatment group will proceed directly into three weeks of baseline and preparation (Days 1 to 18), a 2-dose administration period (Days 22 and 37), integration (Days 23, 30, 38, and 45), the End of Therapy (EOT) visit (Day 52). Participants in the delayed treatment group will wait 8 weeks after enrollment before beginning the study interventions and neuroimaging assessments. As a safety precaution, participants in the delayed treatment group will be assessed weekly via telephone calls or in-person visits during the wait period (i.e., telephone assessments during post-randomization weeks 1, 2, 3, 4, 5, 6, and 7; in-person assessment during post-randomization week 8) to assess suicide risk to determine if intervention is warranted. During week 8, IBS symptoms will also be assessed. At the end of the delay period, all participants in the delayed treatment group will complete the same intervention as the participants in the immediate treatment group.

Validated and commonly used assessment tools will be used to evaluate symptoms at baseline and repeatedly after each session. The weekly average of worst daily pain score and weekly stool frequency and consistency for the 7 days immediately prior to EOT visit will be assessed for change from baseline and at the 3-, 6 , and 12- month follow-up visits (Days 120, 240, 365).

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be 21 to 64 years of age, inclusive, at the time of signing the informed consent form.

Type of Participant and Disease Characteristics

1. Participant has a body mass index (BMI) between 18.5 and 29.9
2. Have a clinical diagnosis of IBS (any subtype) as defined by the Rome IV clinical criteria:
3. Abdominal pain at least 4 days per month over at least 2 months associated with one or more of the following:

   i. Related to defecation ii. A change in frequency of stool iii. A change in form (appearance) of stool iv. After appropriate evaluation, the symptoms cannot be fully explained by another medical condition
4. Have "treatment resistant" IBS (Rajagopalan 1997) by having all of the following:

   1. symptoms for more than 12 months by history
   2. received adequate explanation and reassurance for symptoms as documented by a gastroenterologist in the medical record. This means the patient's primary gastroenterologist will document that they have conducted an evaluation that is within appropriate standards of practice to exclude other medical conditions, and that in their opinion irritable bowel syndrome is the most appropriate diagnosis. The patient's primary gastroenterologist will also document that they have discussed this evaluation and diagnosis with the patient.
   3. tried at least one dietary intervention by history
   4. tried at least one pharmacologic agent for at least six weeks by history
5. Have attempted a gut-brain behavior therapy for at least six weeks by history
6. Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least 2 months prior to screening and is expected to remain stable during participation in the study.
7. Participant must not use tobacco or other nicotine containing products (e.g., vape pens) by history.
8. Participant must be medically stable as determined by screening for medical problems via a personal interview and/or, a medical questionnaire, and an ECG, within 1 month of starting active intervention (performed during screening).
9. Participant must agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea, cola) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of TRP 8802 session days. If the participant does not routinely consume caffeinated beverages, he/she must agree to not do so on the TRP 8802 session day
10. Participant must agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours before and after each TRP 8802 administration. The exception is caffeine.
11. Participant must agree to not take triptan medications (e.g., sumatriptan) within 72 hours before and after each TRP 8802 administration.
12. Participant must agree to not take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours before and after each TRP 8802 administration.
13. Participant must agree to not take any pro re nata (PRN) medications on the mornings of TRP 8802 sessions.
14. Participant must agree that for 7 days before each TRP 8802 session, he/she will refrain from taking any nonprescription medication, cannabis, nutritional supplement, or herbal supplement except when approved by the Principal Investigator. Exceptions will be evaluated by the Principal Investigator and will include acetaminophen, non-steroidal anti-inflammatory drugs, osmotic laxatives, stimulant laxatives, secretagogues such as linaclotide and lubiprostone, birth control, thyroid hormones, and common doses of vitamins and minerals.
15. Participant must have at least a high school level of education or equivalent (e.g., General Educational Development [GED] Test).
16. Participant must demonstrate ability to track abdominal pain and stool frequency and consistency daily in the ePRO system.
17. Participant must demonstrate ability to wear watch with heart rate tracking capability for daily heart rate tracking.
18. Participant must be willing to attempt fMRI scan and EEG. Sex and Contraceptive/Barrier Requirements
19. Contraceptive use by women and men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Adequate birth control methods include intrauterine device, injected/implanted/intravaginal/transdermal hormonal method, oral hormones plus a barrier contraception, abstinence, vasectomized sole partner, or double barrier contraception. Subjects will be excluded if they cannot use highly effective birth control for any reason. If a potential subject lives in an area where local regulations preclude the use of adequate contraception (intrauterine device, injected/implanted/intravaginal/transdermal hormonal method, oral hormones plus a barrier contraception, abstinence, vasectomized sole partner, or double barrier contraception), study enrollment will not be allowed.

    1. If a participant is opting for abstinence as their birth control method, only true/total abstinence is permitted. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), lactational amenorrhea, and withdrawal are not acceptable. Counseling regarding the importance of maintaining abstinence, and the potential risks of exposure to a developing embryo or fetus will be provided during the preparatory sessions during the Preparation 1 session, Integration 1 session, and during Deep Phenotyping 2.
    2. Females of reproductive potential must agree to use effective birth control for the duration of active intervention (defined as the time from the Baseline [deep phenotyping] visit until 6 months and 3 days (for female subjects) after Deep Phenotyping/EOT visit. Female subjects must agree to not donate eggs, or participate in in vitro fertilization for the duration of the recommended contraceptive use of the trial.
    3. Sexually active male participants and/or their female partners must agree to use effective birth control for the duration of active intervention (defined as the time from the Baseline [deep phenotyping] visit until the 3 months and 3 days (for male subjects) after Deep Phenotyping/EOT visit of the male participant. Male participants must also agree not to donate sperm for the duration of active intervention.

    Informed Consent
20. Participant has provided informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Medical Conditions

1. Participant has the following vital sign measurements (taken after 5 minutes of sitting down) during screening visit: SBP>139 mmHg, DBP > 89 mmHg, and/or HR > 90bpm
2. Participant has a history of valvular heart disease reported during screening
3. Participant has a history of pulmonary hypertension reported during screening
4. Participant has moderate to severe hepatic impairment (Child Pugh Class B and C) as determined by presence of ascites or encephalopathy and scoring of albumin, bilirubin, and INR on screening labs
5. Participant has one of the following gastrointestinal medical conditions: inflammatory bowel disease (ulcerative colitis or Crohn's disease), celiac disease, chronic idiopathic constipation, or eosinophilic esophagitis reported during screening
6. Participant has had (within the past 1 year) a cardiovascular condition such as coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged QTc interval (i.e., QTc > 450 msec), artificial heart valve, or transient ischemic attack reported during screening
7. Participant has epilepsy with a history of seizures reported during screening
8. Participant has insulin-dependent diabetes reported during screening
9. Participant is taking an oral hypoglycemic agent and has a history of hypoglycemia.
10. Participant has active auto-immune disease (e.g., lupus, rheumatoid arthritis) reported during screening
11. Participants has any clinically significant lab abnormalities per a complete blood count and metabolic panel (e.g., elevated liver enzymes) at time of screening, and additional screening labs to exclude organic disease within the past two years. Please see screening in Section 4.2. Cutoffs requiring exclusion from the study are listed below:

    Lab Panel Test Cutoff for Exclusion CBC White Blood Cell Count >17 K/uL CBC Hemoglobin <11.5 g/dL CBC Platelets <150 K/uL Metabolic Panel Sodium <130 or >150 Metabolic Panel Potassium <3.2 or > 5.5 Metabolic Panel CO2 <23 or >32 BUN >40 (2X ULN) Creatinine >1.3 Liver Enzymes Direct bilirubin >1.0 Liver Enzymes AST > 80 (2x ULN) Liver Enzymes ALT > 55 (ULN) Clotting Factors INR >4
12. Participant has a current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I or II disorder measured via SCID-5 and SCID-5-PD.
13. Participant has a current or past history (within 1 year) of meeting DSM-5 criteria for a moderate or severe alcohol, tobacco, or other drug use disorder (excluding caffeine) measured via relevant questions from the SCID-5 during screening
14. Participant meets Rome IV criteria for the diagnosis of centrally mediated abdominal pain syndrome (CAPS). Other co-morbid Rome IV diagnoses will not be exclusion criteria.
15. Participant has a history of a medically significant suicide attempt, meaning a suicide attempt leading to an emergency room visit or inpatient hospitalization for any length of time.
16. Participant does not meet institutional guidelines and safety measures for MRI (e.g., has metal in the body or severe claustrophobia) Prior/Concomitant Therapy
17. Participant is taking psychoactive prescription medication (e.g., opioids, tramadol, benzodiazepines) on a regular basis (i.e., more than 2 times a week).
18. Participant is currently taking an antidepressant or neuromodulator, including SSRIs, SNRIs, and TCAs. Participants will also be required to refrain from using antidepressant medications through the completion of primary outcome assessments. Note: if a participant self-initiates a medication taper with the consent and support of their physician, they can re-screen after the appropriate time period.
19. Participant has taken any antidepressant medication for at least 2 weeks (or at least 4 weeks for fluoxetine) prior to the Screening visit.
20. Participant is currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including monoamine oxidase inhibitors (MAOIs). For individuals who have intermittent or PRN use of such medications, TRP 8802 sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
21. Subjects taking serotonin-acting dietary supplements (such as 5-hydroxy-tryptophan or St. John's wort) due to the potential for their interaction with psilocybin and increased safety risks.
22. Subjects taking prohibited medications. The list of prohibited medications includes antihypertensive medications (any ACE-I, ARB, beta blocker, or calcium channel blocker), UGT1A9 or 1A10 inhibitors (e.g., regorafenib, rifampicin, phenytoin, eltrombopag, mefenamic acid, diflunisal, niflumic acid, sorafenib, isavuconazole, deferasiroxor, ginseng) and aldehyde or alcohol dehydrogenase inhibitor (e.g., disulfiram).
23. Participant does not agree to refrain from cannabis use and the use of all other psychoactive medications and drugs of abuse during the study
24. Participant is currently taking prohibited drugs of abuse, including methamphetamine, illicit opioids (e.g., heroin), cocaine, 3,4-methylenedioxymethamphetamine (Ecstasy/Molly), or hallucinogens (e.g., mescaline or peyote).
25. Participant has any use of hallucinogens in the past 6 months or has had a total lifetime hallucinogen use of 10 or more times.
26. Participant tests above 0.02% blood alcohol content on breath alcohol testing and/or positive for cocaine, methamphetamine, or opioids on urine drug testing.
27. Participant has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to TRP 8802.

    Prior/Concurrent Clinical Study Experience
28. Participant is currently in another clinical trial. Diagnostic assessments
29. Participant has a significant suicide risk as defined by:

    1. suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year at Screening or at Baseline; or
    2. suicidal behaviors within the past year; or
    3. clinical assessment of significant suicidal risk during participant interviews Other Exclusions
30. Participant is pregnant (as indicated by a positive urine pregnancy test assessed at Screening and before the TRP 8802 session) or nursing.
31. Participant is a WOCBP and sexually active, or a man and sexually active, and not practicing an effective means of birth control.
32. Participant has a confirmed first- or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I or II disorder.
33. Participant is unable to complete 10/14 days of ePRO tracking during run-in period.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events - Hypertension | Immediately after the intervention
  Incidence of dosing episodes resulting in patient's blood pressure >200 systolic or >110 diastolic for more than 15 minutes (i.e. 4 consecutive readings)
Incidence of Treatment-Emergent Adverse Events - Abuse-Related Psychological Events | Immediately after the intervention
  Presence of "severe" or "extremely severe" (as measured by the Brief Psychiatric Rating Scale [BPRS] hallucinations, psychosis, changes in mood, impaired cognition, attention, psychomotor effects, or inappropriate affect. Note: minimum-maximum scale on BPRS = 0-7, higher score = more severe outcome.
Incidence of Treatment-Emergent Adverse Events - EKG QT Prolongation | Through study completion, an average of 4 months
  Incidence of prolonged QTc (>460ms for women and >450 for men) after receiving at least one dose of psilocybin

SECONDARY OUTCOMES:
Stool consistency | Through study completion, an average of 4 months
  For patients with IBS-Diarrhea (IBS-D), stool consistency as measured by the Bristol Stool Form Scale will be assessed. Patients will answer daily diaries via email about their stooling habits throughout the study. A Stool Consistency Weekly Responder will be defined as a patient who experiences a 50 percent or greater reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline. For patients with IBS-Mixed (IBS-M), bowel function improvement will not be an endpoint. Note: Bristol Stool Form Scale range 1-7, higher number = looser stool.
Stool frequency | Through study completion, an average of 4 months
  For IBS-Constipation (IBS-C), stool frequency as measured by number of complete spontaneous bowel movements (CSBMs) per week, as recorded by daily stool diaries.
Abdominal pain | Through study completion, an average of 4 months
  Patients will answer a daily diary prompt (delivered via email) about their worst daily (in the past 24 hours) abdominal pain. This will be summarized as the weekly average of worst daily abdominal pain score of ≥ 3.0 on a 0 to 10 point scale, with 10 being more severe pain.
Anxiety and depression | Through study completion, an average of 4 months
  Changes in co-morbid anxiety and depression (as measured by Hospital Anxiety and Depression Scale [HADS]). This tool is well-validated in populations with comorbid somatic illness. A HADS anxiety or depression subscore of 11 or greater indicates likely presence of the respective mood disorder. Range 0-21, higher score = more severe.
Severity of IBS | Through study completion, an average of 4 months
  The IBS-Severity Scoring System (IBS-SSS) will be used to generate a summative score incorporating measures of pain, distension, bowel dysfunction and quality of life/global well-being. The maximum (most severe) score is 500, with severe cases scoring > 300. Range 0-500, higher = more severe
GI symptom-specific anxiety | Through study completion, an average of 4 months
  The Visceral Sensitivity Index (VSI) will be used to measure GI-specific anxiety, including the constructs of worry, fear, vigilance, sensitivity, and avoidance. Range 0-75, higher = more severe
Patient Global Impression of Change (PGI-C) | Through study completion, an average of 4 months
  The PGI-C is a questionnaire that gauges the participant's response to medical interventions using a 7-point Likert scale ranging from 1 to 7 with 1 being "very much improved" and 7 being "very much worse" and has been used in many pain clinical trials. Range 1 -7, higher = more severe

OTHER OUTCOMES:
Functional magnetic resonance imaging (fMRI) functional connectivity | Through study completion, an average of 4 months
  Whole-brain images will be acquired to assess for fMRI default mode network (DMN) connectivity. This is presumed to be one way via which psychedelics work. Patients with more centralized pain display increased connectivity between the DMN and the insula, which is diminished with successful treatment. Processed fMRI data will be assessed for seed voxel connectivity between these regions.
Heart rate variability (HRV) | Through study completion, an average of 4 months
  Patients will wear a wristwatch with heart rate tracking and ECG capabilities, from which the metric of heart rate variability will be obtained. IBS patients have measurable autonomic imbalances relative to healthy controls (e.g., diminished parasympathetic modulation during deep breathing and decreased natural logarithm of high frequency power of heart rate variability [LnHF] demonstrating lower vagal tone. Therefore, increased HRV may be a favorable outcome.
Inflammatory biomarkers: High sensitivity C-reactive protein (hsCRP) | Through study completion, an average of 4 months
  Bloodwork will be drawn for inflammatory biomarkers which are known to be involved in the pathogenesis of IBS.
Inflammatory biomarkers: Erythrocyte sedimentation rate (ESR) | Through study completion, an average of 4 months
  Bloodwork will be drawn for inflammatory biomarkers which are known to be involved in the pathogenesis of IBS.
Inflammatory biomarkers: White blood cell (WBC) Count | Through study completion, an average of 4 months
  Bloodwork will be drawn for inflammatory biomarkers which are known to be involved in the pathogenesis of IBS.
Inflammatory biomarkers: Tumor necrosis factor-alpha (TNF-a) | Through study completion, an average of 4 months
  Bloodwork will be drawn for inflammatory biomarkers which are known to be involved in the pathogenesis of IBS.
Inflammatory biomarkers: Interleukin-6 (IL-6) | Through study completion, an average of 4 months
  Bloodwork will be drawn for inflammatory biomarkers which are known to be involved in the pathogenesis of IBS.

CONTACTS AND LOCATIONS:
Overall Officials: Franklin King, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No